CLINICAL TRIAL: NCT00751153
Title: Open Label Phase 4, 48 Week Pilot Study of the Antiviral Efficacy and Tolerability of the Combination of Isentress™ and ReyatazTM When Substituted for Current Antiviral Regimen in Patients With Viral Suppression But Who Are Experiencing Adverse Events Related to Their Current Antiviral Regimen.
Brief Title: Raltegravir and Atazanavir Replacing Current Suppressive Treatment Because of Side Effects in Current Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peter J. Ruane, M.D., Inc. (Other)
Responsible Party: Peter J Ruane, Peter J Ruane MD Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Merck IISP #33040
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2008-10-09 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections
Keywords: drug substitution; Raltegravir; Atazanavir; treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Raltegravir and Atazanavir — Rategravir 400 BID, Atazanavir 400 mg daily

SUMMARY:
Subjects with HIV who have viral suppression on current regimen but also have side effects/intolerance will change their current regimen to a combination of Raltegravir and Atazanavir and be monitored for viral and immunological response and quality of life.

DETAILED DESCRIPTION:
Subjects with intolerance to current regimen will receive Raltegravir 400 mg twice daily and Atazanavir 400 mg daily will be monitored for viralogical and immunological outcomes, changes in lipids, renal and hepatic safety and quality of life.

ELIGIBILITY:
Inclusion Criteria

* History of no PI resistance or antiretroviral failure while receiving a PI.
* On a current antiviral regimen with plasma HIV viral load (VL) < 400 copies/ml for 4 months or longer.
* Intolerance to or toxicity with current or alternative regimen(s) with side effects including but not limited to gastrointestinal, neurological, metabolic, or dysmorphic symptoms and/or dyslipidemia.
* Continuously using the same regimen for 3 months prior to Screening.
* Women of childbearing potential must be willing to use effective method(s) of contraception throughout their study participation and for 30 days following the end of the study (see Section 1.10). -Women who are postmenopausal for at least 2 years, women with total hysterectomy and women with tubal ligation are considered of non-childbearing potential.
* Willing to adhere to the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Use of any drug contraindicated in the current US package insert for Atazanavir or in the investigators brochure for Raltegravir, including PPI inhibitors.
* Use of any investigational drug up to 4 weeks prior to screening.
* Prior or current therapy with Raltegravir.
* Allergy to Raltegravir or Atazanavir
* History of medication non-compliance significant to the study regimen as deemed significant by the investigator.
* Known achlorhydria that would inhibit the absorption of Atazanavir
* Concurrent active chronic Hepatitis B requiring therapy with 3TC, FTC or Tenofovir (entecavir permitted).
* AST or ALT >5 times ULN
* Calculated CrCl < 30 ml/min.
* Female subject who is pregnant or breastfeeding.
* General medical condition that may interfere with the assessments and completion of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the proportion of patients who maintain plasma HIV viral load measurements < 400 copies/ml at week 4, 8, 12, 16, 24, 36 and 48 weeks after switching to Raltegravir and Atazanavir | 48 weeks

SECONDARY OUTCOMES:
Evaluation of the proportion of patients who have plasma HIV viral load measurements <50 copies/ml at week 4, 8, 12, 16, 24, 36 and 48 weeks after switching to Raltegravir and Atazanavir | 48 weeks
Time to virologic failure (defined as 2 consecutive VL measurements > 400 copies/ml on 2 separate clinic visits within 4 weeks) | 48 weeks
Assessment of CD4 cell count changes at 4, 8, 12, 16, 24, 36 and 48 weeks after switching to Raltegravir and Atazanavir | 48 weeks
Assessment of lipid changes after change in regimen | 48 weeks
Determination of incidence, genotypic and phenotypic resistance patterns, in particular to Raltegravir and Atazanavir, in patients in the event of rebound viremia | 48 weeks
Patient adherence to a regimen of Raltegravir and Atazanavir | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Ruane, MB, Principal Investigator — Peter J Ruane MD Inc
Locations (1):
- Medical Practice of Peter Ruane MB, Los Angeles, California, United States